CLINICAL TRIAL: NCT00006342
Title: Analyses of Mutations Associated With Secondary Leukemia or Non-Hodgkin's Lymphoma in Patients Treated for Hodgkin's Disease or Childhood Brain Tumors
Brief Title: Genetic Study in Patients Receiving Treatment for Hodgkin's Disease or Childhood Brain Tumor
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000067681; DUMC-0113-99-1R2; DUMC-IRB-086-97-1; NCI-G00-1840
Record Dates: First submitted 2000-10-04; First posted 2004-05-04 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2013-06

CONDITIONS: Brain and Central Nervous System Tumors; Lymphoma
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; childhood infratentorial ependymoma; childhood low-grade cerebral astrocytoma; childhood supratentorial ependymoma; stage II childhood Hodgkin lymphoma; stage I childhood Hodgkin lymphoma; stage III childhood Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma; childhood high-grade cerebral astrocytoma; untreated childhood brain stem glioma; recurrent childhood brain stem glioma; untreated childhood supratentorial primitive neuroectodermal tumor; recurrent childhood supratentorial primitive neuroectodermal tumor; untreated childhood cerebellar astrocytoma; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; untreated childhood medulloblastoma; recurrent childhood medulloblastoma; newly diagnosed childhood ependymoma; recurrent childhood ependymoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Lymphoma; Hodgkin Disease; Recurrence; Astrocytoma; Medulloblastoma; Familial ependymoma | interventions — Gene Rearrangement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Genetic: chromosomal translocation analysis
Genetic: gene rearrangement analysis
Genetic: mutation analysis

SUMMARY:
RATIONALE: Determination of genetic markers for leukemia or non-Hodgkin's lymphoma that is secondary to Hodgkin's disease and childhood brain tumors may help doctors to identify patients who are at risk for these cancers.

PURPOSE: Clinical trial to determine the presence of certain genes in patients who are receiving treatment for Hodgkin's disease or childhood brain tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the frequency of chromosome 3, 11, and 21 aberrations in peripheral blood lymphocytes (PBL) specifically associated with acute myelogenous leukemia in patients with adult or pediatric Hodgkin's disease treated with radiotherapy and/or chemotherapy. II. Determine the frequency of these aberrations in patients with pediatric central nervous system tumors treated with radiotherapy and/or chemotherapy. III. Determine the glutathione-S-transferase allotype, associated with human toxicological response to carcinogen exposure, for these patients. IV. Determine the frequency of t(14;18) gene rearrangement, associated with deregulation of the bcl-2 proto-oncogene in non-Hodgkin's lymphoma, in PBL of these patients.

OUTLINE: An extra tube of blood is collected before, every 4 weeks during, and every 3 months after radiotherapy and/or chemotherapy. DNA is isolated from the blood sample and the GSTM1, GSTT1, and various cytochrome P (CYP) 450 genotypes are determined by polymerase chain reaction (PCR). Mononuclear leukocytes are analyzed for chromosome aberrations on chromosome numbers 3, 11, and 21. Pretreatment karyotype and frequency of translocations are determined for each patient. Peripheral blood lymphocyte DNA is also examined for t(14;18) gene rearrangements.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of Hodgkin's disease Adult or child OR Diagnosis of primary central nervous system (CNS) malignancy 16 and under Medulloblastoma Ependymoma Brain stem glioma Astrocytoma Primitive neuroectodermal tumor (PNET) Proposed therapy must include external beam radiotherapy and/or chemotherapy

PATIENT CHARACTERISTICS: Age: See Disease Characteristics Any age Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics Surgery: Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 1997-01; Primary Completion 2000-09 (Actual); Study Completion 2001-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward C. Halperin, MD, Study Chair — Duke Cancer Institute
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States